CLINICAL TRIAL: NCT01803659
Title: Effect of Small Daily Doses of B-carotene or Vitamin A on Breast Milk Retinol Concentration in Lactating Filipino Women.
Brief Title: Effect of Small Daily Doses of B-carotene on Breast Milk Retinol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Helen Keller International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6195-2012-01-00-HKI
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Vitamin A Status
Keywords: b-carotene; breastmilk; vitamin A
MeSH Terms: interventions — beta Carotene; retinol palmitate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- b-carotene (Experimental): 600 ug RAE/d as b-carotene, 6 d/wk for 3 weeks
  Interventions: Dietary Supplement: b-carotene
- retinyl palmitate (Active Comparator): 600 ug retinol equivalent/d, 6 d/wk for 3 weeks
  Interventions: Dietary Supplement: retinyl palmitate
- placebo (corn oil) (Placebo Comparator): 0 ug RAE/d as corn oil
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: b-carotene
  Arms: b-carotene
Dietary Supplement: retinyl palmitate
  Arms: retinyl palmitate
Dietary Supplement: placebo
  Arms: placebo (corn oil)

SUMMARY:
The purpose of this pilot study is to determine whether breast milk retinol concentration increases in response to daily supplementation with small amounts of vitamin A (~600 ug RAE/d), as either a b-carotene or retinyl palmitate, 6 d/week for 3 weeks. A secondary purpose is to evaluate sampling methods for collecting breast milk samples in a community setting. The results of this pilot study will allow us to determine whether milk retinol is a useful indicator for evaluating the impact of food-based interventions on the vitamin A status of lactating women.

ELIGIBILITY:
Inclusion Criteria:

* lactating women breastfeeding a single infant 4-12 months of age

Exclusion Criteria:

* chronic disease
* breastfeeding more than one infant
* severe anemia
* signs or symptoms of vitamin A deficiency

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
breast milk retinol concentration | 3 weeks
  breast milk retinol concentration is measured at baseline and after 3 weeks of supplementation with 600 ug RAE/d (as either b-carotene or retinyl palmitate) or 0 ug RAE/d

SECONDARY OUTCOMES:
plasma retinol concentration | 3 weeks
  plasma retinol concentration is measured at baseline and after 3 weeks of supplementation with 600 ug RAE/d (as either b-carotene or retinyl palmitate) or 0 ug RAE/d

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States